CLINICAL TRIAL: NCT02722551
Title: The RELIEF Trial: REduction or eLimination of mItral rEgurgitation in Degenerative or Functional Mitral Regurgitation With the CardiAQ-Edwards™ Transcatheter Mitral Valve
Brief Title: CardiAQ-Edwards™ Transcatheter Mitral Valve Replacement (TMVR) Study
Acronym: RELIEF
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-14
Record Dates: First submitted 2016-03-01; First posted 2016-03-30 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral; Regurgitation; Insufficiency; Degenerative; Functional; Primary; Secondary; Organic; Transcatheter; TMVR; TMVI; Heart valve; Mitral valve; Transapical; Transfemoral; Transeptal; Severe
MeSH Terms: conditions — Mitral Valve Insufficiency; Gastroesophageal Reflux; Neoplasm Metastasis; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the CardiAQ-Edwards™ Transcatheter Mitral Valve (transapical or transseptal delivery)
  Interventions: Device: Transcatheter Mitral Valve Re-placement (TMVR) with the CardiAQ-Edwards™ Transcatheter Mitral Valve

INTERVENTIONS:
Device: Transcatheter Mitral Valve Re-placement (TMVR) with the CardiAQ-Edwards™ Transcatheter Mitral Valve — Replacement of the mitral valve through a transcatheter approach

SUMMARY:
Clinical study to evaluate the safety and performance of the CardiAQ-Edwards™ Transcatheter Mitral Valve

DETAILED DESCRIPTION:
The study is a multi-center, prospective, single-arm, and non-randomized study designed to evaluate the safety and performance of the CardiAQ-Edwards™ Transcatheter Mitral Valve with transapical and transseptal delivery systems in patients with degenerative or functional/ischemic mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* NYHA ≥ II
* Moderate/severe or severe mitral regurgitation
* Prohibitive risk for open-heart surgery
* Meets anatomical criteria

Exclusion Criteria:

* Unsuitable anatomy
* Need for emergent or urgent surgery
* Prior mechanical aortic valve replacement
* Any prior surgical or transcatheter repair (excluding balloon valvuloplasty) or replacement of the mitral valve
* Preexisting device in the left ventricular apex
* Clinically significant, untreated coronary artery disease
* Limited life expectancy (< 12 months)
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2019-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse cardiac and cerebrovascular events | 30 days
  MACCE; all-cause mortality, myocardial infarction, stroke, renal failure, and conversion to surgery per MVARC definitions
Freedom from individual adverse events | 30 days
  % Freedom from individual adverse events

SECONDARY OUTCOMES:
New York Heart Association (NYHA) functional class | 30 days, 3 months, 6 months, 12 months
  Number of patients with improvement in NYHA class
Six minute walk test: | 30 days, 3 months, 6 months, 12 months
  Increase in distance (m) from baseline
Reduction in mitral regurgitation (MR) grade: | 30 days, 3 months, 6 months, 12 months
  Number of patients with reduction in MR grade from baseline
Technical success | 30 days, 3 months, 6 months, 12 months
  Technical success per MVARC criteria (%)
Device success | 30 days, 3 months, 6 months, 12 months
  Device success per MVARC criteria (%)
Procedure success | 30 days, 3 months, 6 months, 12 months
  Procedure success per MVARC criteria (%)
Patient success | 30 days, 3 months, 6 months, 12 months
  Patient success per MVARC criteria (%)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Sondergaard, Principal Investigator — The Rigshospitalet, Copenhagen, Denmark
Locations (15):
- Canada (4):
  - St. Paul's Hospital, University of British Columbia, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Toronto General Hospital, Toronto, Ontario
  - Centre de recherche Institut Universitaire de Cardiologie et de Pneumologie de Québec (CRIUCPQ), Québec
- Rigshospitalet, Copenhagen, Denmark
- Centre Hospitalier Régional Universitaire de Lille, Lille, France
- Germany (5):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Deutsche Herzzentrum Berlin, Berlin
  - Herzzentrum der UniKlinik Köln, Cologne
  - University Heart Centre, Hamburg
  - Leipzig Herzzentrum, Leipzig
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Universita di Roma Tor Vergata, Roma
- Erasmus Medical Centre, Rotterdam, Netherlands
- InselSpital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No